CLINICAL TRIAL: NCT03346850
Title: Comparison Between Gastric and Post Pyloric Tube Feedings in Children With Bronchiolitis Requiring High Flow Nasal Cannula
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of equipoise among enrolling clinicians, as well as emergence of external literature showing safety of nasogastric tube (NGT) feeds.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Raymond Parlar-Chun, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-17-0725
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Enteral Feeding in Bronchiolitis
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- nasogastric tube (NGT) feeding (Active Comparator)
  Interventions: Device: Nasogastric tube (NGT) feeding
- nasoduodenal tube (NDT) feeding (Active Comparator)
  Interventions: Device: Nasoduodenal tube (NDT) feeding

INTERVENTIONS:
Device: Nasogastric tube (NGT) feeding — A nasogastric tube goes from the nose to the stomach.
  Arms: nasogastric tube (NGT) feeding
Device: Nasoduodenal tube (NDT) feeding — A nasoduodenal tube goes from the nose to the duodenum.
  Arms: nasoduodenal tube (NDT) feeding

SUMMARY:
The purpose of the study is to compare two ways (nasogastric tube (NGT) and nasoduodenal tube (NDT)) to provide nutrition to infants admitted to the hospital for viral bronchiolitis and who require high flow nasal cannula therapy.

ELIGIBILITY:
Inclusion Criteria:

- All admitted patients for bronchiolitis requiring high flow nasal cannula therapy at Children's Memorial Hermann

Exclusion Criteria:

* Patients with craniofacial abnormalities that prevent tube placement.
* Patients requiring CPAP and mechanical ventilation are also excluded from the study.
* Patients with past surgeries compromising esophageal sphincter tone such as fundoplication or congenital diaphragmatic hernia surgery are excluded.
* Patients transferred to and from PICU are also excluded from the study.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Parlar-Chun, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Parlar-Chun R, Lafferty-Prather M, Gonzalez V, Pedroza C, Gourishankar A. Protocol: randomised trial to compare nasoduodenal tube and nasogastric tube feeding in infants with bronchiolitis on high-flow nasal cannula; Bronchiolitis and High-flow nasal cannula with Enteral Tube feeding Randomised (BHETR) trial. BMJ Open. 2019 May 5;9(5):e025405. doi: 10.1136/bmjopen-2018-025405. PMID 31061025

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Started | 20 | 20
Completed | 18 | 17
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: days] | 165 (102) | 132 (101) | 148.5 (101.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 4 | 4 | 8
  White | 2 | 3 | 5
  Other | 14 | 13 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Weight [Mean (Standard Deviation); unit: kilograms] | 6.8 (2.6) | 6.1 (2) | 6.45 (2.3)
Number of Participants with Term Gestation [Count of Participants; unit: Participants] | 13 | 14 | 27
Number of Participants with Preterm Gestation [Count of Participants; unit: Participants] | 7 | 6 | 13
Number of participants with spontaneous vaginal delivery (SVD) [Count of Participants; unit: Participants] | 14 | 12 | 26
Number of participants with cesarean delivery (CD) [Count of Participants; unit: Participants] | 6 | 8 | 14
Number of participants with low risk of aspiration [Count of Participants; unit: Participants] | 13 | 14 | 27
Number of participants with high risk of aspiration [Count of Participants; unit: Participants] | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Length of Respiratory Supprt
Time Frame: from the time of hospital admission to discharge (about 6 days)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Number analyzed (Participants) | 20 | 20
hours | 107 (49) | 128 (119)

2. Secondary Outcome: Number of Participants With Emesis
Time Frame: from the time of hospital admission to discharge (about 6 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Number analyzed (Participants) | 20 | 20
Participants | 6 | 1

3. Secondary Outcome: Peak Respiratory Support in Liters Per Minute
Time Frame: from the time of hospital admission to discharge (about 6 days)
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Number analyzed (Participants) | 20 | 20
liters per minute | 8 (1.6) | 7.8 (2.3)

4. Secondary Outcome: Number of Chest X-rays Obtained Among All Participants
Time Frame: from the time of hospital admission to discharge (about 6 days)
Measure: Number; unit: chest x-rays
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Number analyzed (Participants) | 20 | 20
chest x-rays | 31 | 31

5. Secondary Outcome: Number of Participants Who Revisited the Emergency Room (ER)
Time Frame: 7 days after discharge from hospital
Population: 2 in the NGT arm were lost to follow up, and 3 in the NDT arm were lost to follow up; therefore, this data was not collected for these participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Number analyzed (Participants) | 18 | 17
Participants | 1 | 1

6. Secondary Outcome: Number of Participants Who Revisited the Emergency Room (ER)
Time Frame: 30 days after discharge from hospital
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Number analyzed (Participants) | 18 | 17
Participants | 1 | 2

7. Secondary Outcome: Number of Participants Who Were Readmitted to the Hospital
Time Frame: 7 days after discharge from initial hospital visit
Population: 2 in the NGT arm were lost to follow up, and 3 in the NDT arm were lost to follow up; therefore, this data was not collected for these 5 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Number analyzed (Participants) | 18 | 17
Participants | 0 | 1

8. Secondary Outcome: Number of Participants Who Were Readmitted to the Hospital
Time Frame: 30 days after discharge from initial hospital visit
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
Number analyzed (Participants) | 18 | 17
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From the time of enrollment to discharge (about 6 days)
Arm/Group | Nasogastric Tube (NGT) Feeding | Nasoduodenal Tube (NDT) Feeding
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasogastric Tube (NGT) Feeding (N=20) | Nasoduodenal Tube (NDT) Feeding (N=20)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasogastric Tube (NGT) Feeding (N=20) | Nasoduodenal Tube (NDT) Feeding (N=20)
nose bleed (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT03346850/Prot_SAP_000.pdf